CLINICAL TRIAL: NCT02471118
Title: Osteoarthritis of the Knee, Inflammation, and the Effect of Adalimumab (OKINADA): A Randomized Placebo-controlled Trial
Brief Title: Osteoarthritis of the Knee, Inflammation, and the Effect of Adalimumab (OKINADA)
Acronym: OKINADA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: CARE ARTHRITIS LTD. (Industry)
Collaborators: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IMM 11-0024
Record Dates: First submitted 2015-02-24; First posted 2015-06-15 (Estimated); Last update posted 2021-10-27 (Actual); Status verified 2021-10

CONDITIONS: Osteoarthritis, Knee
Keywords: Inflammatory Type
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Adalimumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1st 50 subjects to Enter the Study (Experimental): At Baseline, subjects will be randomized (1:1) to receive study drug (Adalimumab or placebo). The study drug will be provided as a subcutaneous injection (pre-filled syringe) either Adalimumab (ADA) 40 mg/0.8 mL,every other week (EOW) or matching placebo for Adalimumab every other week for 16 weeks. Efficacy will be assessed at Week 16 while the safety of the study drug will be monitored throughout the study.
  At Week 16 all subjects will begin to receive open label ADA 40 mg EOW and will continue to receive open label ADA up to Week 50. An End of Study visit will be done at Week 52. A Telephone Follow-up will be done at Week 62 to review Adverse Events and Concomitant Medications.
  Interventions: Drug: Adalimumab 40 mg; Drug: Placebo
- 2nd group of 50 subjects (Experimental): At Baseline, subjects will be randomized (1:1) to receive either adalimumab 40 mg every other week or placebo for 16 weeks. All subjects will begin to receive open label adalimumab 40 mg every other week from week 16-week 30, with An End of Study visit at Week 32. A Telephone Follow-up will be done at Week 42 to review Adverse Events and Concomitant Medications.
  Interventions: Drug: Adalimumab 40 mg; Drug: Placebo

INTERVENTIONS:
Drug: Adalimumab 40 mg — Adalimumab will be self-administered via subcutaneous (SC) injection
  Other Names: Humira
Drug: Placebo — Placebo will be self-administered via subcutaneous (SC) injection

SUMMARY:
This is a Canadian randomized, double-blind, placebo-controlled, multicenter study designed to evaluate the clinical efficacy and safety of adalimumab versus placebo when used to treat subjects with a diagnosis of osteoarthritis of the knee, and with clinical features of inflammation, whose pain persists despite receiving maximum tolerated doses of conventional therapy.

DETAILED DESCRIPTION:
This is a Canadian randomized, double-blind, placebo-controlled, multicenter study designed to evaluate the clinical efficacy and safety of adalimumab versus placebo when used to treat subjects with a diagnosis of osteoarthritis of the knee, and with clinical features of inflammation, whose pain persists despite receiving maximum tolerated doses of conventional therapy. A total of 100 subjects will be entered into the study.

Subjects will be randomized (1:1) at baseline to receive either adalimumab 40 mg every other week or placebo for 16 weeks. The study drug will be self-administered via subcutaneous injection. Efficacy will be assessed at week 16 while the safety of the study drug will be monitored throughout the study. At week 16 all subjects will begin to receive open label adalimumab 40 mg every other week.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 40 years of age
2. If female, subject is either not of childbearing potential, defined as postmenopausal for at least 1 year or surgically sterile (bilateral tubal ligation, bilateral oophorectomy or hysterectomy), or is of childbearing potential and practicing methods of birth control.
3. If female and of childbearing potential, serum pregnancy results must be negative at Screening
4. Has a diagnosis of Osteoarthritis (OA) of the index knee according to American College of Rheumatology (ACR) criteria, including radiological evidence of OA (Kellgren-Lawrence grades 2 or 3).
5. Subject has had knee pain for at least 1 month prior to the Screening Visit.
6. Subject has had knee pain that has persisted despite conventional treatment, defined as any one of the following medications taken for at least 1 month in the past:

   * acetaminophen (2- 4 grams per day)
   * therapeutic dose range of an NSAID
   * acetaminophen/codeine combination (i.e. Tylenol No. 2, 3, 4) taken at least 3 times daily.
7. Has a pain score of ≥ 4 (0-10 NRS) in the index (more symptomatic) knee at Screening and Baseline.
8. If the subject is taking Analgesic/NSAIDs, then the Analgesic/NSAIDs has been stable for 14 days prior to the Baseline visit.
9. Has clinical evidence of a knee effusion in the index (more symptomatic) knee at Screening and Baseline.
10. Able and willing to self-administer SC injections or has available qualified person(s) to administer SC injections.
11. Has voluntarily signed and dated an approved informed consent form prior to any study-specific procedures.

Exclusion Criteria:

1. Has a history of an allergic reaction or significant sensitivity to constituents of adalimumab.
2. Has other bone and articular diseases (antecedents and/or current signs) such as chondrocalcinosis, Paget's disease of the ipsilateral limb to the target knee, rheumatoid arthritis, aseptic osteonecrosis, gout, septic arthritis, ochronosis, acromegaly, haemochromatosis, Wilson's disease, osteochondromatosis, seronegative spondylo-arthropathy, mixed connective tissue disease, collagen vascular disease, psoriasis, inflammatory bowel disease.
3. Subject has a BMI over 40.
4. Planned/anticipated surgery of the index knee during the study period.
5. Already scheduled for any surgery during the time of the study or within 70 days after the end of treatment.
6. Prior arthroscopic or open surgery of the index knee within 12 months of Baseline.
7. Has a history of cancer or lymphoproliferative disease other than: Successfully and completely treated cervical dysplasia, with no recurrence within the last five years, Basal or Squamous Cell Carcinoma that has been adequately treated or excised.
8. Has had prior treatment with intravenous (IV) immunoglobulin or any investigational agent within 30 days or 5 half-lives of the agent from Baseline, whichever is longer.
9. History of neurologic symptoms suggestive of central nervous system (CNS) demyelinating disease (e.g. multiple sclerosis).
10. History of uncontrolled diabetes, unstable ischemic heart disease, active congestive heart failure, New York Heart Association (NHYA) III, IV, inflammatory bowel disease, active peptic ulcer disease, recent stroke (within 12 weeks of Screening), or any other condition, which in the opinion of the investigator, would put the patient at risk by participating in the study.
11. Has concurrent local or systemic infection that would preclude the use of adalimumab.
12. Has had a persistent or severe infection(s) requiring hospitalization or treatment with IV antibiotics within 30 days, or oral antibiotics within 14 days, prior to Baseline.
13. History of active tuberculosis or listeriosis, or other infections suggestive of significant or profound immunosuppression, such as Pneumocystis carinii, aspergillosis or other systemic protozoal or fungal infections.
14. Has latent TB (positive purified protein derivative (PPD) skin test, two-step PPD when applicable, and chest X-ray indicative of TB) or has other risk factors for the activation of latent TB, e.g. previous exposure to TB, and has not initiated TB prophylaxis prior to the first adalimumab treatment.
15. Will be excluded if the Chest x-ray is found to have changes indicative of old healed tuberculous lesion (e.g. calcified nodule, fibrotic scar, apical or basilar pleural thickening etc.).
16. Has a positive serology for Hepatitis B or Hepatitis C that indicates active infection.
17. Has a history of positive HIV status.
18. Currently taking or likely to begin anti-retroviral therapy at any time during the course of the study.
19. Female subject is pregnant or breast-feeding.
20. Has a history of clinically significant drug or alcohol abuse in the last year, prior to Screening.
21. Subject, in the opinion of the principal investigator, is unlikely to comply with the study protocol or is unsuitable for any other reason.

Treatment-Related Exclusion Criteria

1. Subject has received intra-articular injections of steroid and/or hyaluronate compounds into the index knee within 12 weeks prior to Baseline.
2. Subjects using injectable corticosteroids for any medical condition (intra-articular/soft tissue injections are allowed, but not in the target knee).
3. Subjects using indomethacin or oral steroids.
4. Subjects taking glucosamine and/or chondroitin at screening must discontinue or remain on a stable dose, unmodified if at all possible for the entire duration of the study.
5. If treatment for osteoarthritis (NSAID) or osteoporosis (bisphosphonates, selective estrogen receptor modulators) is necessary, it will have to be continued, unmodified if at all possible for the entire duration of the study. If the subject does not wish to continue them during the study, they must be stopped 14 days prior to the Baseline visit.
6. Subjects who have used compounds containing non-approved agents for arthritis or agents claiming to possess disease/structure-modifying properties in the 14 days prior to the Baseline visit (see exception above).
7. Subjects who require acetaminophen at daily doses > 4000 mg (4 g) on a regular basis.
8. Subjects who are taking lithium carbonate, phenytoin or anticoagulants (with the exception of aspirin up to a maximum daily dose of 325 mg).
9. Subjects who use calcitonin.
10. Subjects who use immunosuppressive drugs. Subjects that are using methotrexate or hydroxychloroquine must withdraw treatment 1 month prior to baseline, to be eligible to enter the study.
11. Topical analgesics and NSAID's cannot be used on the target knee within the 48 hours before each study visit.
12. No new physical modalities of treatment can be introduced and subject must maintain normal activity during the study.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2021-03 (Actual); Study Completion 2021-03 (Actual)

PRIMARY OUTCOMES:
Primary Endpoint: the percentage of subjects achieving an Osteoarthritis Research Society International/Outcome Measures in Rheumatology Clinical trials (OARSI/OMERACT) response at Week 16 | 16 weeks
  The primary efficacy outcome measure will be the percentage of subjects achieving an OARSI/OMERACT response at Week 16.

SECONDARY OUTCOMES:
Secondary endpoint Knee Injury and Osteoarthritis Outcome (KOOS) composite pain score at 16 weeks. | 16 weeks
  1. KOOS composite pain score at 16 weeks.
Secondary endpoint KOOS composite pain 20/50 response rates | 16 weeks
  2. KOOS composite pain 20/50 response rates, i.e., the percentages of subjects showing ≥ 20% and ≥ 50% improvements from baseline in KOOS composite pain scores in the index knee at 16 weeks.
Secondary Endpoint KOOS activities of daily living score | 16 Weeks
  3. KOOS activities of daily living score at 16 weeks.
Secondary Endpoint KOOS symptoms score | 16 weeks
  4. KOOS symptoms score at 16 weeks.
Secondary Endpoint KOOS sport and recreation function score | 16 weeks
  5. KOOS sport and recreation function score at 16 weeks.
Secondary Endpoint KOOS knee-related quality of life score | 16 weeks
  6. KOOS knee-related quality of life score at 16 weeks.
Secondary Endpoint Patient global assessment of disease status score | 16 weeks
  7. Patient global assessment of disease status score at 16 weeks.
Secondary Endpoint Investigator global assessment of disease status score | 16 Weeks
  8. Investigator global assessment of disease status score at 16 weeks.
Secondary Endpoint Physical assessment of Target Joint | 16 weeks
  9. Physical assessment of Target Joint at 16 weeks.
Secondary Endpoint Expanded Target Joint Assessment score | 16 weeks
  10. Expanded Target Joint Assessment score at 16 weeks.
Secondary Endpoint Average weekly consumption of analgesic medications | 16 weeks
  11. Average weekly consumption of analgesic medications over 16 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Walter P Maksymowych, MD, FRCPC, Study Director — CARE ARTHRITIS LTD.
Locations (7):
- Canada (7):
  - Division of Rheumatology, University of Alberta Hospital, Edmonton, Alberta
  - Western University, London, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - A.M.I.R., Montreal, Quebec
  - GRMO Inc., Québec, Quebec
  - CHUS Hotel-Dieu, Sherbrooke, Quebec
  - Polmed Research Inc., Saskatoon, Saskatchewan

REFERENCES:
- [Background] 1. National Advisory Council on Aging and Public Health Agency of Canada, Division of Aging and Seniors. Musculoskeletal disorders such as arthritis and osteoporosis [Online]. Available at http://www.naca-ccnta.ca/vignette/vig69_e.htm#69. 2. Malemud CJ. Cytokines as therapeutic targets for osteoarthritis, BioDrugs 2004;18:23- 35. 3. Abramson SB, Yazici Y. Biologics in development for rheumatoid arthritis: Relevance to osteoarthritis. 4. Pelletier JP, Martel-Pelletier J, Abramson SB.Osteoarthritis, an inflammatory disease: potential implication for the selection of new therapeutic targets. Arthritis Rheum. 2001;44:1237-1247. 5. Felson DT, McLaughlin S, Goggins J, LaValley MP, Gale ME, Totterman S, Li W, Hill C, Gale D: Bone marrow edema and its relation to progression of knee osteoarthritis. Ann Intern Med 2003, 139:330-336. 6. Hunter DJ, Zhang Y, Niu J, Goggins J, Amin S, LaValley MP, Guermazi A, Genant H, Gale D, Felson DT: Increase in bone marrow lesions associated with cartilage loss: a longitudinal magnetic resonance imaging study of knee osteoarthritis. Arthritis Rheum 2006, 54:1529-1535. 7. Kornaat PR, Kloppenburg M, Sharma R, Botha-Scheepers SA, Le Graverand MP, Coene LN, Bloem JL, Watt I: Bone marrow edema-like lesions change in volume in the majority of patients with osteoarthritis; associations with clinical features. Eur Radiol 2007, 17:3073-3078. More references available